CLINICAL TRIAL: NCT03602313
Title: Biomechanical Gait Analysis in Patients Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-40
Record Dates: First submitted 2018-05-04; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: CVA (Cerebrovascular Accident); Stroke
Keywords: Body Weight Support
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to 1 of 2 groups for the duration of the study.
Who Masked: Investigator
Masking Description: Investigators were blinded to the study intervention. Data collection was performed at a separate location than the primary intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Gait Training (Active Comparator): The Traditional Gait Training group will receive gait training as presently performed without additional modalities.
  Interventions: Other: Traditional Gait Training
- Body Weight Support Training (Experimental): The Body Weight Support group will received body weight support gait training in lieu of traditional gait training.
  Interventions: Device: Body Weight Support Gait Training

INTERVENTIONS:
Device: Body Weight Support Gait Training
  Other Names: BSWTT, LiteGait
  Arms: Body Weight Support Training
Other: Traditional Gait Training
  Other Names: Overground
  Arms: Traditional Gait Training

SUMMARY:
Randomized trial of patients with cerebrovascular accident (CVA) receiving traditional and body weight supported (BWS) gait training. Participants are enrolled and randomized upon entry into acute care and gait is evaluated within 48 hours of discharge from the rehabilitation hospital. Gait analysis is used to determine which of the two groups achieved gait parameters most similar to the normal gait of an age-matched population.

DETAILED DESCRIPTION:
Potential participants are identified upon admission to acute care post cerebrovascular accident (CVA) and screened for inclusion. Informed consent is obtained from the patient and/or designee. Demographic information is obtained from the medical record, the patient and/or designee by the clinical coordinator. The participant is randomized into traditional gait training group or body weight support (BWS) group. The participant receives the required amount of physical therapy as directed by clinicians at the acute care facility and accrediting agencies.

The traditional gait training group will receive gait training as presently performed without additional modalities. The BWS group will received BWS gait training in lieu of traditional gait training. Participants will be treated in in-patient rehabilitation for a duration as determined by the clinical team; thus, the overall duration of care may be variable between participants. Time spent in gait training activities for both groups will be tracked by both service unit and by time (minutes).

Within 48 hours of discharge from the acute care facility, the participant will be transported to a separate site for kinematic gait analysis using a marker based motion capture system.

The procedure for gait analysis is as follows:

1. Investigators will place reflective markers on the following areas using non-latex adhesive tape: top of the shoulders, bony part of the pelvis on the front and back, hips, front of the thighs, outside of the knees, front of the shins, outside of the ankles, first and fifth toes, and back of each heel.
2. The participant will walk across the room in the gait analysis lab no more than 20 times at his/her choice of pace while the camera system records gait parameters and kinematics. He/she will be allowed to rest as needed during the data collection.
3. The reflective markers and adhesive tape will be removed and the participant thanked for his/her participation.

ELIGIBILITY:
Inclusion Criteria:

* Current in-patient in acute care for Cerebrovascular accident (CVA),
* Unilateral CVA affecting at least the lower limb, and
* Medically stable as determined by the rehabilitation physician.

Exclusion Criteria:

* Previous (more than 1) CVA with residual lower limb deficit, and
* Any lower extremity pathology on the affected side other than the effects of the CVA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12-06 (Actual); Primary Completion 2015-09-17 (Actual); Study Completion 2015-09-17 (Actual)

PRIMARY OUTCOMES:
Gait Speed | Collected in one 1-hour session after the patient has completed acute rehabilitation, approximately 21 days.
  Velocity of center of mass of the participant.
Step Length | Collected in one 1-hour session after the patient has completed acute rehabilitation, approximately 21 days.
  Difference in position between the feet at heel strike, in the direction of forward motion.
Step Width | Collected in one 1-hour session after the patient has completed acute rehabilitation, approximately 21 days.
  Difference in position between the feet at heel strike, in the direction normal to the direction of forward motion.
Step Asymmetry | Collected in one 1-hour session after the patient has completed acute rehabilitation, approximately 21 days.
  The ratio of the difference of left and right step length over the stride length.

SECONDARY OUTCOMES:
Gait Units | Measured at discharge, approximately 21 days
  Measure of the quantity of therapy received during the duration of care.
Functional Independence Measure (FIM) | Admission of the FIM is completed within 72 hours of the start of a rehabilitation, and within 75 hours of discharge, approximately 21 days
  A 17 items survey of patient independence in 2 domains, motor and cognition. It is used as a basic indicator of patient disability.
Length of Stay | Approximately 21 days. Determined by the study clinicians based on severity of disability and rate of progress.
  Total duration of care at the acute rehabilitation facility.

CONTACTS AND LOCATIONS:
Overall Officials: Derek J Lura, PhD, Principal Investigator — Florida Gulf Coast University